CLINICAL TRIAL: NCT01495546
Title: Randomized Comparison of Quality of Life and Functional Patients Undergoing Total Hip Replacement Uncemented. Load Early X Load Late
Brief Title: Total Hip Arthroplasty (THA): Early Load Versus Load Late
Acronym: Latearly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Gisele Pucci Mantelli, Physiotherapist, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CAPPesq0303
Record Dates: First submitted 2011-12-12; First posted 2011-12-20 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Primary Total Hip Arthroplasty
Keywords: total hip arthroplasty; THA; prosthesis type Lepine
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early loading (Experimental)
  Interventions: Other: Early loading
- late loading (Active Comparator)
  Interventions: Other: Late loading

INTERVENTIONS:
Other: Early loading — Patients stepping down immediately after THA
  Arms: Early loading
Other: Late loading — Patients stepping down after three weeks of HTA
  Arms: late loading

SUMMARY:
In Brazil, several hip surgeries performed, especially total knee arthroplasty, which represents 1.5 million procedures (Penedo, New, 2007). The rehabilitation of these individuals is slow with respect to the march because it requires an aid and not to use the operated leg as support for three weeks, according to conventional methods. After the third week, the support becomes part and after that period (sixth week), the support becomes total. Therefore, and in order to provide better quality of life, the goal of this work is to compare the march in 40 patients divided into two groups of 20 subjects each. In the control group, the treatment approach is the traditional, i.e., without immediate loading, while the other charge will be applied immediately in the operated limb. In order to verify the possible gain in the quality of life of these patients, the SF-36 will be applied. The march will be assessed with the Time Up and Go test and the force platform and the Harris Hip score analyze the function of the hip. Individuals will receive such care at the Institute of Orthopedics and Traumatology, Hospital das Clinicas, Faculty of Medicine, University of São Paulo (IOT - HC - USP). The results of comparisons between the two groups and the clinical findings obtained will be subjected to appropriate statistical tests, guided by the principles of evidence-based clinical practice, seeking to facilitate and improve the lives of these individuals so they can move freely.

ELIGIBILITY:
Inclusion Criteria:

* Patients served by the institution with THA without cement;
* BMI less than 40, ie, present in most class II obesity;
* Patients with diseases such as osteoarthritis and osteonecrosis of the femoral head;
* Absence of systemic involvement;
* Patients with prosthetic type Lépine.

Exclusion Criteria:

* Bilateral arthroplasty;
* Partial arthroplasty;
* Arthroplasties for review;
* Cemented arthroplasties;
* Surgical complications.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Recovery time after THA | Until 6 weeks
  Patients will be evaluated in the following periods: THA pre-surgery, the third day post-surgery THA, third and sixth week post-surgery THA, third and sixth months after surgery THA

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Orthopedics and Traumatology, Hospital das Clinicas, Faculty of Medicine, University of Sao Paulo, São Paulo, São Paulo, Brazil